CLINICAL TRIAL: NCT07229521
Title: Effects of Nattokinase on Cardiovascular Disease Risk Factors, Gut Microbiota, Sleeping and Cognitive Function in Patients With Risk of Metabolic Syndrome Along With Sleeping Disorder.
Brief Title: Effects of Nattokinase on Cardiovascular Risk, Gut Microbiota, Sleep, and Cognition in Metabolic Syndrome With Sleep Disorders.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N202412072
Record Dates: First submitted 2025-04-08; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-02

CONDITIONS: Metabolic Syndrome; Sleeping Disorders
MeSH Terms: conditions — Metabolic Syndrome; Parasomnias | interventions — nattokinase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: nattokinase (Experimental): Dietary supplement: nattokinase (containing nattokinase 3000FU per capsule) This group will be given supplements for 12 weeks.
  Interventions: Dietary Supplement: Nattokinase
- Placebo Comparator: placebo (Placebo Comparator): Placebo treatment (identical capsules containing Microcrystalline Cellulose)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Nattokinase — Participants will be divided into a placebo group and an experimental group. The experimental period was divided into two phases (12 weeks for each) and a 2-week washout period. In the first phase, 2 nattokinase capsules were given each day (each capsule contained nattokinase 3000FU, 2 capsules per day). After 12 weeks, a 2-week washout period was entered, and the second phase was entered for a crossover trial.
  Arms: Experimental: nattokinase
Other: Placebo — Participants will be divided into a placebo group and an experimental group. The experimental period was divided into two phases (12 weeks for each) and a 2-week washout period. In the first phase, 2 placebo capsules were given each day (each capsule contained Microcrystalline Cellulose, 2 capsules per day). After 12 weeks, a 2-week washout period was entered, and the second phase was entered for a crossover trial.
  Arms: Placebo Comparator: placebo

SUMMARY:
Nattokinase has been confirmed by many experiments to have a thrombolytic effect, but there are currently very few studies on nattokinase's effect on gut microbiota, sleeping status, and age-related cognitive function. Therefore, this study intends to explore the effect of nattokinase on cardiovascular disease risk factors, intestinal microbiota, sleep status and cognitive function in patients with metabolic syndrome risk and sleep disorders. This study will be a double-blind, self-control, placebo, crossover trial, and recruit 70-80 participants over 18 years old, and have risk of metabolic syndrome and sleep disorders. They will be divided into a placebo group and an experimental group. The experimental period was divided into two phases (12 weeks for each) and a 2-week washout period. In the first phase, 2 placebo or nattokinase capsules were given each day (each capsule contained nattokinase 3000FU, 2 capsules per day). After 12 weeks, a 2-week washout period was entered, and the second phase was entered for a crossover trial. At the 0th and 12th weeks of each stage, body position, blood pressure, blood biochemical values, sleep quality questionnaire, and cognitive function questionnaire will be measured, and feces will be collected for bacterial analysis. In addition, to improve the compliance of the trial, it is planned to ask the subjects to return for a follow-up visit in the 6th week of each phase, and to measure the subject's body composition and blood pressure. This study expects that daily supplementation of 2 nattokinase capsules for 12 weeks can improve cardiovascular risk factors, sleep quality and cognitive function, while also maintaining healthy intestinal flora.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old
2. Meet the criteria of MetS: meet at least two of the following four items will be recognized as at risk of metabolic syndrome:

   1. Abdominal obesity: Male≧90cm (35 inches); Female≧80cm (31inches)
   2. High blood pressure: Systolic blood pressure≧120mmHg or diastolic blood pressure≧80mmHg
   3. High fasting blood glucose: Fasting blood glucose≧100mg/dL
   4. Dyslipidemia: High fasting triglycerides (≧150mg/dL) or low high-density lipoprotein cholesterol (HDL-C) (<40mg/dL for male, <50mg/dL for female)
3. The Apnea Hypopnea Index (AHI) was diagnosed by overnight multi-channel sleep physiology examination (Polysomnography, PSG) or Home Sleep Apnea Test (HSAT) to be between 5 and 30, indicating mild or moderate sleep apnea.
4. No major mental illness or obvious symptoms of anxiety or depression
5. No combination with other primary sleep diseases

Exclusion Criteria:

1. Body mass index (BMI) >30 kg/m^2
2. Chronic diseases: abnormal liver and kidney function, abnormal gastrointestinal function, cardiovascular disease, high blood pressure, diabetes mellitus, and hyperlipidemia, etc.
3. Participants requiring medication for conditions not specified in exclusion criterion (2), who are unable to maintain a stable treatment regimen throughout the trial
4. Malignant tumors
5. Pregnancy or breastfeeding
6. Person expected to perform the surgery.
7. Those who have participated in other clinical trials in the past 28 days.
8. May be allergic to the ingredients in the test materials, or take drugs or dietary supplements that may affect the test results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2026-12-11 (Estimated); Study Completion 2027-02-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline The Pittsburgh Sleep Quality Index (PSQI) at 3 months | At 0th week, and 12th week for each of the two phases.
  PSQI is used to evaluate sleeping quality. A self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval.
Change from Baseline Insomnia Severity Scale at 3 months | At 0th week, and 12th week for each of the two phases.
  ISI is a simple self-assessment questionnaire for evaluating the severity of insomnia, assessing the severity of insomnia over the past two weeks in the study participants.
Change from Baseline Epworth Sleepiness Scale (ESS) at 3 months | At 0th week, and 12th week for each of the two phases.
  ESS is a self-administered questionnaire, and is used to assess the "daytime sleepiness" of the patients.
Change from Baseline Patient Health Questionnaire at 3 months | At 0th week, and 12th week for each of the two phases.
  PHQ-9 is a widely used tool for assessing depressive symptoms in both clinical and research settings, evaluating the severity of depressive symptoms over the past two weeks through 9 questions.
Change from Baseline Generalized Anxiety Disorder at 3 months | At 0th week, and 12th week for each of the two phases.
  GAD-7 is a brief self-report scale specifically designed to assess the frequency and severity of anxiety symptoms over the past two weeks.
Change from Baseline Oguri-Shirakawa-Azumi Sleep Inventory MA version at 3 months | At 0th week, and 12th week for each of the two phases.
  OSA Sleep Inventory MA version is a psychological measurement tool suitable for clinical settings and for middle-aged and elderly individuals who are unable to appropriately respond to multiple-choice questions, used to assess an individual's self-evaluation of sleep upon waking.
Change from Baseline The Cambridge Neuropsychological Test Automated Battery at 3 months | At 0th week, and 12th week for each of the two phases.
  CANTAB (Cambridge Neuropsychological Test Automated Battery) is a computerized cognitive function testing system developed by the University of Cambridge, This study will use the preclinical dementia test battery recommended by CANTAB. This test battery has been proven to have better sensitivity and discriminative ability compared to traditional assessment methods including ADAS-cog and MMSE, and can detect cognitive function changes in the short to medium term.
  The overall assessment includes the following 7 subtests:
  1. Motor Screening Task (MOT)
  2. Reaction Time (RTI)
  3. Paired Associates Learning (PAL)
  4. Spatial Working Memory (SWM)
  5. Pattern Recognition Memory (PRM)
  6. Delayed Matching to Sample (DMS)
  7. Rapid Visual Information Processing (RVP)

SECONDARY OUTCOMES:
Anthropometric Assessment | At 0th week, 6th week, and 12th week for each of the two phases.
  body weight (kg)
Anthropometric Assessment | At 0th week, 6th week, and 12th week for each of the two phases.
  Body fat mass (%/kg)
Anthropometric Assessment | At 0th week, 6th week, and 12th week for each of the two phases.
  Skeletal muscle mass (%/kg)
Blood pressure | At 0th week, 6th week, and 12th week for each of the two phases.
  blood pressure (mmHg)
Liver Function | At 0th week, and 12th week for each of the two phases.
  Serum AST (U/L)
Liver Function | At 0th week, and 12th week for each of the two phases.
  Serum ALT (U/L)
Kidney Function | At 0th week, and 12th week for each of the two phases.
  Serum BUN (mg/dL)
Kidney Function | At 0th week, and 12th week for each of the two phases.
  Creatinine (mg/dL)
Kidney Function | At 0th week, and 12th week for each of the two phases.
  eGFR (mL/min)
Kidney Function | At 0th week, and 12th week for each of the two phases.
  uric acid (mg/dL)
Lipid Profile | At 0th week, and 12th week for each of the two phases.
  Serum HDL-C (mg/dL)
Lipid Profile | At 0th week, and 12th week for each of the two phases.
  Serum LDL-C (mg/dL)
Lipid Profile | At 0th week, and 12th week for each of the two phases.
  Serum triglyceride (mg/dL)
Lipid Profile | At 0th week, and 12th week for each of the two phases.
  Serum total cholesterol (mg/dL)
Hematology | At 0th week, and 12th week for each of the two phases.
  Complete Blood Count
Antioxidative Status | At 0th week, and 12th week for each of the two phases.
  Concentration of thiobarbituric acid-reactive substance
Antioxidative Status | At 0th week, and 12th week for each of the two phases.
  Glutathione/oxidized glutathione ratio.
Fecal Microbiota | At 0th week, and 12th week for each of the two phases.
  Using 16S rRNA and next-generation sequencing to analyze gut microbiota composition.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan